CLINICAL TRIAL: NCT06416956
Title: Baby-CINO: CaffeINe Treatment Optimisation in Premature Infants
Acronym: Baby-CINO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: PID17161; 23/SC/0397 (Other: Research Ethics Committee)
Record Dates: First submitted 2023-12-15; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2023-12

CONDITIONS: Infant,Premature; Caffeine
MeSH Terms: conditions — Premature Birth | interventions — Caffeine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preterm infant: Preterm infants receiving caffeine (prescribed clinically) will be studied
  Interventions: Drug: Caffeine

INTERVENTIONS:
Drug: Caffeine — We will record infant's brain activity and vital signs when caffeine dose is changed or caffeine treatment is stopped. The decision to change dose/stop treatment will be made by the clinical team as part of routine care. No changes in caffeine treatment will be carried out solely for research purposes.

SUMMARY:
This study investigates how brain activity and breathing changes in premature babies when their dose of caffeine treatment is changed or stopped. The study will assess premature babies receiving caffeine treatment as part of their clinical care. Brain activity will be recorded just before caffeine dose is changed and again two days afterwards. Breathing and other 'vital signs' (breathing rate, heart rate, oxygen saturation) will be recorded from the baby's monitor between the recordings of brain activity and for up to two weeks afterwards.

ELIGIBILITY:
Inclusion Criteria:

* Born to a mother aged 16 or over
* Admitted to the Newborn Care Unit, John Radcliffe Hospital
* Born prematurely (before 37 weeks' gestation)
* Parent given informed written consent
* Receiving caffeine citrate

Exclusion Criteria:

* Known chromosomal abnormality or life-threatening congenital abnormality
* Severe hypoxic insult at birth
* Intraventricular haemorrhage grade III or IV or other severe neurological pathology

Max Age: 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All participants will be inpatients on the Newborn Care Unit and born prematurely (before 37 weeks gestation)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Respiration | From baseline to two days later
  Change in respiratory dynamics between baseline (time at which caffeine dose is changed/treatment ends) and approximately 2 days later
Brain activity | From baseline to two days later
  Change in EEG activity between baseline (time at which caffeine dose is changed/treatment ends) and approximately 2 days later

SECONDARY OUTCOMES:
Heart rate | From baseline to two days later
  Change in heart rate between baseline (time at which caffeine dose is changed/treatment ends) and approximately 2 days later
Oxygen saturation | From baseline to two days later
  Change in oxygen saturation between baseline (time at which caffeine dose is changed/treatment ends) and approximately 2 days later

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Hartley, Principal Investigator — University of Oxford
Locations (1):
- Newborn Care Unit, John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided